CLINICAL TRIAL: NCT07163143
Title: Optimal Treatment Duration for Radiographically Apparent, Bacteriologically Unconfirmed TB, Identified Through Active Case Finding
Brief Title: Optimal Treatment Duration for Radiographically Apparent, Bacteriologically Unconfirmed TB, Identified Through Active Case Finding (RADIO-TB Trial)
Acronym: RADIO-TB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National University of Medical Sciences, Pakistan (Other); Aurum Institute (Other); Biomedical Research and Training Institute, Zimbabwe (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); KTH Royal Institute of Technology (Other); London School of Hygiene and Tropical Medicine (Other); Wits Health Consortium (Pty) Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 314897/Z/24/Z
Record Dates: First submitted 2025-08-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis (TB)
Keywords: Treatment duration; Radiographically apparent TB; Bacteriologically unconfirmed TB; Response over continuous intervention (ROCI); Active case finding; Asymptomatic; Subclinical; Chest X-ray; Screening; Computer Aided Detection (CAD)
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Protons; Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment (Active Comparator): Immediate start of 24 weeks (approx. 6 months) TB treatment comprised of 8 weeks (approx. 2 months) isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE) followed by 16 weeks (approx. 4 months) of isoniazid and rifampicin (4HR) - 2HRZE/4HR
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)
- Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment (Experimental): Immediate start of 20 weeks (approx. 5 months) TB treatment comprised of 8 weeks (approx. 2 months) isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE) followed by 12 weeks (approx. 3 months) of isoniazid and rifampicin (3HR) - 2HRZE/3HR
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)
- Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment (Experimental): Immediate start of 16 weeks (approx. 4 months) TB treatment comprised of 8 weeks (approx. 2 months) isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE) followed by 8 weeks (approx. 2 months) of isoniazid and rifampicin (2HR) - 2HRZE/2HR
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)
- Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment (Experimental): Immediate start of 12 weeks (approx. 6 months) TB treatment comprised of 8 weeks (approx. 2 months) isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE) followed by 4 weeks (approx. 1 month) of isoniazid and rifampicin (1HR) - 2HRZE/1HR
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)
- Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment (Experimental): Immediate start of 8 weeks (approx. 2 months) TB treatment comprised of isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE)
  Interventions: Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Pyrazinamide (Z); Drug: Ethambutol (E)
- Arm F. No initial treatment, deferred if progression. (No Intervention): No initial treatment - if during close follow-up there is bacteriological confirmation and/or clinical/radiological progression, to start 24 weeks (approx. 6 months) TB treatment - 2HRZE/4HR

INTERVENTIONS:
Drug: Isoniazid (H) — H, weight based, 150-375mg
  Arms: Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment; Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment; Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment; Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment; Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment
Drug: Rifampicin (R) — R, weight based, 300-750mg
  Arms: Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment; Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment; Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment; Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment; Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment
Drug: Pyrazinamide (Z) — Z, weight based, 800-2000mg
  Arms: Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment; Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment; Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment; Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment; Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment
Drug: Ethambutol (E) — E weight based, 550-1375mg
  Arms: Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment; Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment; Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment; Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment; Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment

SUMMARY:
People living in high TB burden communities who undergo active case finding for TB may have chest X-ray changes suggestive of TB but their sputum test can be negative for the TB bacteria or they are unable to provide a sputum sample. This means they have bacteriologically unconfirmed TB. These individuals often have minimal or no symptoms and face uncertainty in clinical management-either receiving full 24-weeks TB treatment or often being discharged without treatment, risking loss to follow-up.

The RADIO-TB trial aims to address the following main questions in relation to people with bacteriologically unconfirmed TB.

1. What is the risk of progression if treatment is not immediately started but there is close and careful follow-up over 78 weeks?
2. If treatment is started immediately what is the shortest duration of TB treatment that is as effective as the standard 24-week TB treatment?
3. Are there better tests to confirm TB than the current routinely used, sputum-based tests?
4. What is the cost effectiveness of different treatment strategies and what might the impact on transmission be within communities?

Participants in the trial will be randomized into six groups: five receiving immediate standard TB treatment of varying durations (8 to 24 weeks), and one receiving deferred treatment with close monitoring. Deferred treatment will be initiated only if clinical deterioration occurs or TB is later confirmed. Participants will be closely followed for 78 weeks with at least 11 clinic visits.

DETAILED DESCRIPTION:
Increasingly, countries are adopting community-based chest X-ray (CXR) screening strategies to identify people with TB at an early stage, often before they have symptoms. However, a significant proportion of individuals with radiographic abnormalities suggestive of TB are not bacteriologically confirmed due to limitations in sputum-based diagnostics or inability to produce sputum. These individuals are often diagnosed with "bacteriologically unconfirmed TB," and there is currently no consensus on how best to manage them.

The RADIO-TB trial is a multi-country, multi-arm, phase 3 clinical trial designed to address this critical evidence gap. The trial aims to determine the optimal treatment duration for individuals with radiographic evidence of TB who do not have bacteriological confirmation and are identified through active case finding (ACF) using CXR and computer-aided detection (CAD) software. The study is being conducted in South Africa, Zimbabwe, and Pakistan. Recruitment for the trial will be conducted alongside existing programatic CXR-based TB ACF activity taking place in these countries.

RADIO-TB uses a pragmatic, open-label, randomized design with six parallel arms. Participants are randomized to one of the following 6 arms in a ratio 1:1:1:1:1:2.

Arm A. Immediate start of 24 weeks (approx. 6 months) TB treatment comprised of 8 weeks (approx. 2 months) isoniazid, rifampicin, pyrazinamide and ethambutol (2HRZE) followed by 16 weeks (approx. 4 months) of isoniazid and rifampicin (4HR) - 2HRZE/4HR (control-A).

Arm B. Immediate start of 20 weeks (approx. 5 months) TB treatment - 2HRZE/3HR. Arm C. Immediate start of 16 weeks (approx. 4 months) TB treatment - 2HRZE/2HR. Arm D. Immediate start of 12 weeks (approx. 3 months) TB treatment - 2HRZE/1HR. Arm E. Immediate start of 8 weeks (approx. 2 months) TB treatment - 2HRZE. Arm F. No initial treatment, deferred if progression - if during close follow-up there is bacteriological confirmation and/or clinical/radiological progression, to start 24 weeks (approx. 6 months) TB treatment - 2HRZE/4HR (control-F).

The trial employs a Response Over Continuous Intervention (ROCI) design, which allows for the estimation and modelling of the duration-response curve and a more precise and efficient identification of the shortest non-inferior treatment duration compared to the standard 24-week regimen. The study hypothesis is that those with radiographically apparent, bacteriologically unconfirmed TB identified through ACF, immediate TB treatment with duration that is 8 weeks or longer, but less than 24 weeks, will be: (A) Non-inferior to treatment of 24 weeks duration (Arm A) at a 5% non-inferiority margin and (B) Superior to no initial treatment (Arm F) to prevent unfavourable TB outcomes.

The trial will enrol 784 participants aged 16 years and older who have undergone CXR-based TB ACF locally and found to have a CAD score above a locally defined threshold for TB investigation and either sputum negative by a WHO-approved rapid molecular test for TB or are unable to produce sputum. Key exclusion criteria are: a history of prior pulmonary TB, evidence of extra-pulmonary TB, clinical indication for immediate full-course treatment or an alternative cause for the CXR abnormalities more likely than TB. People who are HIV-infected will be eligible if their CD4 count is ≥200/mm3 and they on established on anti-retroviral therapy (ART). The CAD software used for screening will be those used locally in the existing ACF programmes according to international recommendation and national approvals. At the end of the study CXR will be re-analysed for all available CAD software to aid generalisability of findings.

All participants will undergo comprehensive baseline assessments, including clinical evaluation, induced sputum culture, blood and respiratory sampling for novel diagnostics. They are followed for 78 weeks with scheduled clinical evaluations, repeat chest X-ray, repeat microbiological testing, and quality-of-life assessments. Where necessary participants will be investigated for conditions other than TB.

The primary outcome measure for the trial is the proportion with unfavourable outcomes defined as requiring initiation of TB treatment after the week 0 visit for either bacteriologically confirmed TB or clinical/radiological progression without bacteriological confirmation. The trial also evaluates safety, tolerability of treatment; the impact on lung function, chest X-ray changes and quality of life; the frequency and timing of diagnoses other than TB; and the development of drug resistance. In addition, the study includes ancillary components to (1) assess the cost-effectiveness of different treatment strategies, (2) model the impact of different strategies on TB transmission and (3) evaluate novel diagnostic tools that may improve the early identification and confirmation of TB.

The RADIO-TB trial is sponsored by University College London (UCL) and funded by the Wellcome Trust. It is coordinated by the UCL Institute of Clinical Trials and Methodology (ICTM) in collaboration with national TB programs, academic institutions, and community partners in the participating countries. The trial incorporates robust patient and public involvement (PPI) mechanisms to ensure that the research is aligned with community priorities and that findings are disseminated in accessible and impactful ways.

By generating high-quality evidence on the optimal management of bacteriologically unconfirmed TB, the RADIO-TB trial aims to inform national and international TB treatment guidelines. The results will support more individualised and evidence-based approaches to TB care, improve patient outcomes, and contribute to global efforts to end the TB epidemic.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥16 years old on day of randomisation
2. ≥25kg in weight on day of randomisation
3. Participation in community or facility-based active case finding for TB by CXR
4. Digital CXR with Computer Aided Detection software score above threshold for sputum investigation for Mtb according to local guidance ≤21 days prior to randomisation
5. Attempted sputum collection for testing by WHO approved rapid molecular test for Mtb at active case finding and at screening

Exclusion Criteria:

1. Sputum sample from active case finding or screening confirmed as positive for Mtb by WHO approved rapid molecular test for Mtb
2. Previous history of pulmonary TB
3. TB preventive therapy taken within the last 6 months
4. >1 dose of treatment with anti-tuberculous activity taken in the 21 days prior to randomisation
5. HIV infected, unless CD4 ≥200 cells/mm3 and on anti-retroviral therapy for at least 8 weeks
6. Pregnancy (confirmed by high sensitivity urine test)
7. Contraindication to study drug
8. Investigator concern for potential extra-pulmonary TB with the exceptions of (a) intrathoracic lymphadenopathy; and/or (b) small pleural effusion of limited extent, neither felt to require invasive diagnostic sampling
9. CXR changes considered more likely to relate to a condition other than untreated TB by investigator
10. Investigator assessment of an immediate requirement for full 24-weeks standard TB treatment
11. Investigator assessment of unacceptable risks to potential participant from study entry
12. No fixed home address
13. Unable to participate in the full duration of study follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 784 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an unfavourable TB outcome | Over 78 weeks post-randomisation
  Unfavourable outcome = requiring initiation of TB treatment after the week 0 visit for either bacteriologically confirmed TB or clinical/radiological progression without bacteriological confirmation

SECONDARY OUTCOMES:
Time to (re-)treatment | Over 78 weeks post-randomisation
Proportion of participants with bacteriological confirmation for Mtb | Over 78 weeks post-randomisation
Proportion of participants initiated on TB treatment for symptomatic TB | Over 78 weeks post-randomisation
Computer Aided Detection (CAD) software score (TB related) | At weeks 8, 36 and 72
  Higher score indicates a higher probability of TB related abnormality.
Forced expiratory volume in 1 second (FEV1) | At 72 weeks
  Lung function test determined by spirometry
Forced vital capacity (FVC) | At 72 weeks
  Lung function test determined by spirometry
FEV1/FVC ratio | At 72 weeks
  Lung function test determined by spirometry
Total time on TB treatment | Over 78 weeks
Number Needed to Treat to prevent unfavourable outcome | Over 78 weeks
All-cause mortality | Over 78 weeks
Proportion of participants experiencing Grade 2/3/4 Adverse Events (AE) (and the subset which are treatment emergent) according to DAIDS criteria | Over 24 and 78 weeks
Proportion of participants experiencing Serious Adverse Events | Over 24 and 78 weeks
Proportion of participants experiencing Hepatotoxicity AE of Special Interest | Over 24 and 78 weeks
Proportion of participants permanently stopping treatment due to an AE of any grade (AESI) | Over 78 weeks
Proportion of participants with final diagnosis of baseline CXR abnormality as non-TB | Over 78 weeks
Time to non-TB diagnosis | Over 78 weeks
Proportion who develop isoniazid and/or rifampicin resistant TB | Over 78 weeks
EuroQol Visual Analogue Scale score | Over 72 weeks
  Scaled - 0 (worst imaginable health) to 100 (best imaginable health)
Short Form 36 (SF-36) score | At weeks 0, 8, 16, 24, 48, 72
  36 item questionnaire evaluating 8 health domains. Domains are scored 0 (worse health) to 100 (better health).
Chronic Obstructive Pulmonary Disease Assessment Test (CAT) score | At 72 weeks
  8 item questionnaire. Individual question scores are summed to provide a total score ranging from 0 to 40. A higher score indicates a greater impact of lung condition on their health and daily life.

OTHER OUTCOMES:
Change in Computer Aided Detection software scores (multi-domain) | Over 72 weeks
  Will include TB-related scores provided by software and other abnormality scores.
Extent of TB related symptoms determined by NCI-PRO-CTCAE custom survey | Over 24 and 72 weeks
Extent of treatment tolerability determined by NCI-PRO-CTCAE custom survey | Over 24 and 72 weeks
Quality adjusted Time without Symptoms and Toxicity (Q-TWiST) | Over 78 weeks
Extent of treatment acceptance determined by the PROMIS Scale v1.0 Medication Adherence questionnaire | Over 78 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- National University of Medical Sciences, Islamabad, Pakistan
- South Africa (2):
  - Clinical HIV Research Unit, Wits Health Consortium, Johannesburg
  - The Aurum Institute, Johannesburg
- Bulawayo City Health, Bulawayo, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Plan to upload IPD to public repository e.g. WHO IPD or TB-PACTS
Supporting Information: Study Protocol
Time Frame: After primary publication (est Q4 2029)
Access Criteria: Via application to the IPD repository